CLINICAL TRIAL: NCT00002432
Title: An Open Study of Foscarnet Treatment of CMV-Retinitis in AIDS Patients
Brief Title: A Study of Foscarnet in the Treatment of Cytomegalovirus (CMV) of the Eyes in Patients With AIDS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Astra USA (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Purpose: Treatment
Other Study IDs: 020E; 89-FOS-06
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1990-07

CONDITIONS: Cytomegalovirus Retinitis; HIV Infections
Keywords: Retinitis; AIDS-Related Opportunistic Infections; Foscarnet; Cytomegalovirus Infections; Acquired Immunodeficiency Syndrome
MeSH Terms: conditions — Cytomegalovirus Retinitis; HIV Infections; Retinitis; AIDS-Related Opportunistic Infections; Cytomegalovirus Infections; Acquired Immunodeficiency Syndrome | interventions — Foscarnet

INTERVENTIONS:
Drug: Foscarnet sodium

SUMMARY:
To evaluate the safety and efficacy of foscarnet induction therapy for treatment of AIDS patients experiencing their first episode of cytomegalovirus (CMV) retinitis. To evaluate the safety and efficacy of foscarnet maintenance therapy for treatment of AIDS patients experiencing CMV retinitis.

ELIGIBILITY:
Inclusion Criteria

Prior Medication:

Allowed:

* Ganciclovir (DHPG).

Exclusion Criteria

Co-existing Condition:

Patients with the following are excluded:

* Any clinically significant pulmonary or neurologic impairment (e.g., patients who are intubated or comatose).
* Corneal, lens, or vitreous opacification which precludes examination of the fundi, or evidence of tuberculotic, diabetic, and/or hypertensive retinopathy.
* Known allergy to foscarnet.

Concurrent Medication:

Excluded:

* Nephrotoxic drugs.
* Acyclovir.

Patients with the following are excluded:

* Any clinically significant pulmonary or neurologic impairment (e.g., patients who are intubated or comatose).
* Corneal, lens, or vitreous opacification which precludes examination of the fundi, or evidence of tuberculotic, diabetic, and/or hypertensive retinopathy.
* Known allergy to foscarnet.

Prior Medication:

Excluded within 7 days of study entry:

* Immunomodulators.
* Biologic response modifiers.
* Investigational agents (other than ganciclovir).

Patients with AIDS as defined by the CDC, with manifest first episode cytomegalovirus (CMV) retinitis as identified by its characteristic ophthalmoscopic appearance and verified by fundus photography.

* Patients must be able to give informed consent.
* Patients who enter the study because of ganciclovir toxicity will have received ganciclovir therapy which resulted in either absolute neutrophil count falling to < 750 cells/mm3 or platelet count falling to < 50000 platelets/mm3 on two separate occasions during either:
* A ganciclovir induction regimen of 7.5 mg (or more)/kg/day in divided doses.
* A maintenance regimen of 5 mg (or more)/kg/day as a single daily dose.
* Patients who enter the study because of ganciclovir treatment failure will meet one of the following criteria:
* CMV retinitis progression has occurred either 1) at the end of a 10 - 21 day induction course of ganciclovir (7.5 - 10 mg/kg/day in divided doses) or 2) during the first 28 days of maintenance ganciclovir therapy (5 mg (or more)/kg/day, at least 5 days/week) where maintenance therapy began within 1 week of completing induction therapy.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (1):
- Davies Med Ctr, San Francisco, California, United States

REFERENCES:
- [Background] Leonard L, Lippe M, Follansbee S, Drennan D, Karol C. An open study of foscarnet treatment of cytomegalovirus (CMV) retinitis in AIDS patients. Int Conf AIDS. 1990 Jun 20-23;6(1):231 (abstract no ThB436)